CLINICAL TRIAL: NCT04076787
Title: The Effect of Vascular Endothelial Growth Factor Receptor (VEGFR) Tyrosine Kinase Inhibitors (TKI) on Clinical Outcomes Among Patients With Metastatic Renal Cell Carcinoma (mRCC) Who Received First-Line Sunitinib in the International mRCC Database Consortium (IMDC) Based on Prognostic Risk Score
Brief Title: Clinical Outcomes for Patients With Renal Cell Carcinoma Who Received First-Line Sunitinib
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) (Other); Analysis Group, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181229
Record Dates: First submitted 2019-08-30; First posted 2019-09-03 (Actual); Results first posted 2019-10-10 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2021-02

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Vascular endothelial growth factor (VEGF); Sunitinib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Favorable IMDC risk group: The cohort of mRCC patients receiving sunitinib as first-line treatment and classified as favorable IMDC risk group for having 0 individual risk factor
  Interventions: Drug: Sunitinib
- Intermediate IMDC risk group: The cohort of mRCC patients receiving sunitinib as first-line treatment and classified as intermediate IMDC risk group for having 1 or 2 individual risk factors
  Interventions: Drug: Sunitinib
- Poor IMDC risk group: The cohort of mRCC patients receiving sunitinib as first-line treatment and classified as poor IMDC risk group for having 3 or more individual risk factors
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — patients who received sunitinib as first line therapy for mRCC

SUMMARY:
This is a retrospective, longitudinal cohort study that assessed clinical outcomes of patients with metastatic renal cell carcinoma (mRCC) who received sunitinib as first-line treatment.

DETAILED DESCRIPTION:
Clear cell mRCC patients who initiated sunitinib as first-line treatment between 2010 and 2018 were identified from the IMDC database. Patients were classified as favorable, intermediate, or poor prognostic risk group according to IMDC criteria. Overall survival, time to treatment discontinuation, and physician-assessed tumor response were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with mRCC
* Initiated treatment post mRCC diagnosis and received sunitinib as first-line therapy
* Age 18 years or over at the time of mRCC diagnosis
* Actively treated at an IMDC clinical center

Exclusion Criteria:

* Initiated first line sunitinib treatment before 2010
* Had non-clear cell mRCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with clear cell mRCC at age 18 or older who initiated sunitinib as first-line treatment between 2010 and 2018
Sampling Method: Non-Probability Sample
Enrollment: 1769 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-09-02 (Actual); Study Completion 2018-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A6181229

RESULTS

PARTICIPANT FLOW:
Recruitment Details: International metastatic renal cell carcinoma database consortium (IMDC) real-world database was used to collect the data from the medical charts of adult participants with clear metastatic renal cell carcinoma (mRCC), who received first-line sunitinib therapy in a real-world setting, from January 2010 to February 2018.
Groups:
- IMDC Prognostic Risk Group: Favorable: Participants with clear mRCC, who received first-line sunitinib therapy in a real-world setting, from January 2010 to February 2018 and were stratified IMDC prognostic risk group as favorable survival group (with no IMDC risk factor).
- IMDC Prognostic Risk Group: Intermediate: Participants with clear mRCC, who received first-line sunitinib therapy in a real-world setting, from January 2010 to February 2018 and were stratified IMDC prognostic risk group as intermediate survival group (with 1 or 2 IMDC risk factor).
- IMDC Prognostic Risk Group: Poor: Participants with clear mRCC, who received first-line sunitinib therapy in a real-world setting, from January 2010 to February 2018 and were stratified IMDC prognostic risk group as poor survival group (with 3 or more than 3 IMDC risk factor).
Period: Overall Study
Arm/Group | IMDC Prognostic Risk Group: Favorable | IMDC Prognostic Risk Group: Intermediate | IMDC Prognostic Risk Group: Poor
Started | 318 | 1031 | 420
Completed | 318 | 1031 | 420
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all adult participants with clear mRCC treated with first-line sunitinib.
Groups:
- Total: Total of all reporting groups
Arm/Group | IMDC Prognostic Risk Group: Favorable | IMDC Prognostic Risk Group: Intermediate | IMDC Prognostic Risk Group: Poor | Total
Number analyzed (Participants) | 318 | 1031 | 420 | 1769
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (9.6) | 62.9 (10.2) | 62.6 (9.6) | 63.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 259 | 117 | 460
  Male | 234 | 772 | 303 | 1309
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 183 | 505 | 209 | 897
  Non-white | 34 | 119 | 46 | 199
  Not reported | 101 | 407 | 165 | 673

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time between index date and death due to any cause or end of data availability. The index date was defined as the date of initiation of first-line sunitinib therapy.
Time Frame: 60 months
Population: Analysis population included all adult participants with clear mRCC treated with first-line sunitinib. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMDC Prognostic Risk Group: Favorable | IMDC Prognostic Risk Group: Intermediate | IMDC Prognostic Risk Group: Poor
Number analyzed (Participants) | 117 | 553 | 327
months | 52.1 [43.4 to 61.2] | 31.5 [28.9 to 33.9] | 9.8 [8.3 to 11.4]

2. Primary Outcome: Time to First-Line Sunitinib Treatment Discontinuation
Description: Time to treatment discontinuation was defined as the time between index date and either discontinuation of first-line sunitinib therapy due to any reason including disease progression, death, toxicity, both disease progression and toxicity, other or end of data availability. The index date was defined as the date of initiation of first-line sunitinib therapy.
Time Frame: 60 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMDC Prognostic Risk Group: Favorable | IMDC Prognostic Risk Group: Intermediate | IMDC Prognostic Risk Group: Poor
Number analyzed (Participants) | 244 | 884 | 383
months | 15.0 [12.4 to 17.3] | 8.5 [8.0 to 9.5] | 4.2 [3.4 to 4.9]

3. Primary Outcome: Number of Participants Who Discontinued First-Line Sunitinib Treatment
Description: In this outcome measure, participants who discontinued treatment due to any reason like disease progression, death, toxicity, both disease progression and toxicity, other or end of data availability are reported.
Time Frame: 60 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IMDC Prognostic Risk Group: Favorable | IMDC Prognostic Risk Group: Intermediate | IMDC Prognostic Risk Group: Poor
Number analyzed (Participants) | 157 | 536 | 206
Participants
  Disease progression | 91 | 316 | 122
  Toxicity | 52 | 141 | 42
  Other reasons | 11 | 54 | 22
  Death | 2 | 17 | 13
  Disease progression and toxicity | 1 | 8 | 7

4. Primary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR are defined as the disappearance of all lesions (target and/or non target). Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter. PR are those with at least 30 percent (%) decrease in the sum of diameters of the target lesions taking as a reference the baseline sum diameters.
Time Frame: 60 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | IMDC Prognostic Risk Group: Favorable | IMDC Prognostic Risk Group: Intermediate | IMDC Prognostic Risk Group: Poor
Number analyzed (Participants) | 288 | 902 | 350
percentage of participants | 38.5 | 34.6 | 21.7

5. Primary Outcome: Percentage of Participants With Progressive Disease
Description: Progressive disease (PD) was defined as an increase in visible disease. According to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) progressive disease: - at least a 20% increase in the sum of diameters of target lesions taking as reference the smallest sum on the study. This includes the baseline sum if that is the smallest on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: 60 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | IMDC Prognostic Risk Group: Favorable | IMDC Prognostic Risk Group: Intermediate | IMDC Prognostic Risk Group: Poor
Number analyzed (Participants) | 288 | 902 | 350
percentage of participants | 16.3 | 27.1 | 46.0

6. Primary Outcome: Percentage of Participants With Stable Disease
Description: Stable disease was defined as no change in size of visible disease. According to Response Evaluation Criteria in Solid Tumors (RECIST 1.1), stable disease neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive disease: - at least a 20% increase in the sum of diameters of target lesions taking as reference the smallest sum on the study. PR are those with at least 30 percent (%) decrease in the sum of diameters of the target lesions taking as a reference the baseline sum diameters.
Time Frame: 60 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | IMDC Prognostic Risk Group: Favorable | IMDC Prognostic Risk Group: Intermediate | IMDC Prognostic Risk Group: Poor
Number analyzed (Participants) | 288 | 902 | 350
percentage of participants | 45.1 | 38.4 | 32.3

ADVERSE EVENTS:
Time Frame: Not applicable as safety data were not collected during the study
Description: Safety data were not planned to be collected during the study.
Arm/Group | IMDC Prognostic Risk Group: Favorable | IMDC Prognostic Risk Group: Intermediate | IMDC Prognostic Risk Group: Poor
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT04076787/Prot_SAP_000.pdf